CLINICAL TRIAL: NCT06934330
Title: Effect of Tao Calligraphy Meditation and Energized Water on Depression Randomized Control Cross-over Study
Brief Title: Effect of Tao Calligraphy Meditation and Energized Water on Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sha Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00050084
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Unipolar Depression
Keywords: Unipolar Depression; Well-being; SF 36 Quality of life questionnaire; PHQ-9 questionnaire; Tao Calligraphy; Healing Art; Chinese Calligraphy; BAI-21 Beckman Anxiety Inventory
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: The study will be performed as a 3-month randomized control cross-over study. The participants will be adults (19 years and older). New participants may enter the study at any time and will be randomized into either the practice group or the control group.
  The practice group will start practices at the baseline zero time point and will stop their practices at the 6-weeks time point. The control group will crossover to the practice group at the 6-weeks time point and will stop practices at the 12-weeks time point.
  The study will evaluate the effects of mindfulness practice using these standardized questionnaires:
  * the SF-36 Quality of Life questionnaire,
  * the PHQ-9 Questionnaire and
  * the BAI-21 Beckman Anxiety Inventory
  All participants will complete the set of all three questionnaires upon entry into the study - the baseline zero time point; and again, at the 6-weeks and the 12-weeks time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Group (Experimental): The Practice group will start practices at baseline zero time point and will stop practices after six weeks at 6-weeks time point. Participants in the Practice group will practice Mindfulness practice with Calligraphy at least 30 minutes daily and drink about 1 litre of Energized water daily for six weeks. All participants in the Practice group will complete the set of all three questionnaires upon entry into the study - at the baseline zero time point; at the 6-weeks time point and at the 12-weeks time point.
  Interventions: Behavioral: Mindfulness practice with Tao Art (Calligraphy and Song Greatest Love); Other: Drinking Energized water
- Control Group (No Intervention): The Control group will crossover to become Practice group at the 6-weeks time point. Participants will start practices at the 6-weeks time point and will stop practices after six weeks at 12-weeks time point.
  All participants in Control Group will complete the set of all three questionnaires upon entry into the study at Baseline time point; at 6-weeks time point and at 12-weeks time point.

INTERVENTIONS:
Behavioral: Mindfulness practice with Tao Art (Calligraphy and Song Greatest Love) — During mindfulness practice with Tao Art (Calligraphy and Song Greatest Love), participants will repeatedly trace the lines of calligraphy with fingers while listening to, singing, or chanting with Tao Song. This enables them to achieve deep concentration, while maintaining fully alert state. The practice can be done in sitting or standing, depending on the health status and age and will last 30 minutes and is done daily for six weeks.
  Arms: Practice Group
Other: Drinking Energized water — Participants will drink energized water from a bottle that received subtle energy transmission. They will replenish water daily and activate the transmission in the bottle to energize the water. Participants will drink about 1 litre of energized water a day for six weeks.
  Arms: Practice Group

SUMMARY:
The goal of this controlled randomized clinical study is to learn if a Tao Calligraphy Mindfulness and Energized water Practice works to improve Unipolar Depression. The main questions it aims to answer are:

* Does Tao Calligraphy Mindfulness practice and drinking Energized water improve the subjective symptoms of Unipolar Depression in adults?
* Does Tao Calligraphy Mindfulness practice and drinking Energized water improve the clinical symptoms and signs of Unipolar Depression in adults?
* Will any improvement in the John Ware's SF-36 Quality of Life questionnaire, in the Patient Health Questionnaire (PHQ) -9 and in the Beckman Anxiety Inventory (BAI) -21 in adults be statistically significant? Investigators will compare the values of these three scales at the beginning of the mindfulness and energized water practices to their values at six weeks of practice and control groups.

Participants will:

* be randomized into practice and control groups
* complete the set of three questionnaires upon entry into the study - (the baseline or zero time point; at the 6-weeks time point, and at the 12-weeks time point
* practice the mindfulness techniques with Tao Calligraphy for a minimum of thirty minutes daily and energized water practice for a minimum of five minutes daily.

DETAILED DESCRIPTION:
Objective

The goal of this study is to measure the positive effects of a unique form of mindfulness practice that involves engaging with Tao art (tracing the Tao Calligraphy "Greatest Love" while listening to or singing the Tao Music or Tao Song "Greatest love") combined with energized water drinking on human adult well-being and depression symptoms and signs. Investigators will study the impact of this Tao art mindfulness practice on three standard research instruments: the John Ware's SF-36 Quality of Life questionnaire, the PHQ-9 questionnaire and the BAI-21 Beckman Anxiety Inventory

Hypotheses

The research hypotheses are that individuals with unipolar depression who receive energy transmission (blessing) for their affliction, who will regularly practice meditations with Tao Calligraphy and drink energized water will report:

1. a decrease in the symptoms of their illness as perceived subjectively.
2. an improvement of the clinical status of their illness, as observed by their clinicians.
3. improvement of well-being or clinical status as measured by standardized scientific questionnaire (s).

For statistical analysis of scores obtained from questionnaires, the Anova and regression analysis will be used to evaluate the null hypothesis. The p value will represent how unlikely the observed data would be if the null hypothesis were actually true and investigators will use them to reach conclusions. The confidence level is set at 95% and if we receive p < 0.05, then results are considered statistically significant. The correlation coefficient will be used to determine any correlation between various factors (e.g. effects of age, sex, length, and frequency of mindfulness practices and other) on outcome and regression analysis will be used to determine the relation of independent and dependent variables.

Background and Theoretical Framework

Depression is a mental disorder characterized by a depressed mood, lack of interest, decreased concentration, decreased self-esteem, increased fatigue, reduced activity, feelings of worthlessness, drive reduction for longer periods of time and suicidal thoughts. Depression affects a person's thoughts, behaviour, feelings and sense of well-being. Depression is one of the most common mental disorders, affecting more than 300 million people of all ages globally, and is now the leading cause of disability. Depression is a major contributor to mortality, morbidity, disability, and economic costs in the United States. Centre for Disease Control and Prevention (CDC) analyzed 2020 Behavioral Risk Factor Surveillance System (BRFSS) data to estimate the national, state-level, and county-level prevalence of U.S. adults aged ≥18 years self-reporting a lifetime diagnosis of depression (referred to as depression). During 2020, the age-standardized prevalence of depression among adults was 18.5%.

Mindfulness meditation-based therapies are being increasingly used as interventions for psychiatric disorders. Mindfulness refers to a state of awareness that arises from paying attention to the present moment, without judgment, whereas meditation refers to a practice or technique that can cultivate mindfulness, inner peace, and more. Mindfulness practices are often synonymous with meditation, and the terms are often used interchangeably.

Mindfulness practices have become increasingly popular as complementary therapeutic strategies for a variety of medical and psychiatric conditions. Likewise, mindfulness and meditation practices have been shown to increase self-compassion and improve memory and emotional regulation. In a comprehensive meta-analysis of 209 studies, the authors concluded that mindfulness-based therapy was effective for many types of psychological problems, while being especially good for reducing anxiety, depression, and stress. In another overall review of mindfulness-based interventions, they were found to be effective for many common and diverse mental, physical, and social conditions.

In recent decades, mindfulness and meditation practices and programs have become increasingly commonplace for stress management and reduction because they are effective. It is no wonder that mindfulness-based meditation practices lead to greater mental, physical, and psychological well-being, with one of the key mechanisms for such outcomes being their effect on the regulation or reduction of stress.

Besides mindfulness and meditation practices, the interest in the application of the arts for public health and well-being has also grown in recent years. Self-expression through art or engaging with different forms of art has been found to be helpful for many health conditions, and doctors in the United Kingdom have started prescribing "the arts" to treat or positively influence many kinds of health conditions.

Some forms of art are also meditative and contemplative, and many can be readily transformed into such a process. The mindfulness-based meditation being explored in this research rests in part on the benefits of music, singing or chanting, and calligraphy tracing (in particular, tracing a unique form of Chinese calligraphy).

Chinese calligraphic writing is a dynamic process that uses an ink-laden brush to create defined configurations of characters. Revered as one of the most important art forms in China, as a mindfulness practice, it has also been shown to help reduce stress and improve mental well-being. The practice of Chinese calligraphy writing facilitates the development of concentration, creativity, and relaxation, which can lead to a more peaceful mental state. Studies in the medical field have confirmed its significant effects on psychosomatic conditions, post-traumatic hyper-arousal symptoms, hypertension, and type 2 diabetes. Other research publications have shown how it can improve cognitive function in the elderly, improve neuropsychiatric symptoms, and reduce stress. In one case, a man who was in a coma for two years awakened and continued to improve after his medical team took his hand and helped him to trace calligraphy daily with his finger.

This research will explore the effects of a unique mindfulness-based meditation that combines tracing the Tao Calligraphy "Greatest Love" while listening to, singing, or chanting the Tao Song "Greatest Love" and drinking energized water. Investigators will study its effect upon general well-being and upon specific depressive symptoms.

Tao Calligraphy is based on a unique branch of Chinese calligraphy known as Yi Bi Zi, which applies one-stroke writing. Every character is written with one continuous stroke of the brush, with the brush always in contact with the paper.

In a unique style of moving meditation, participants will focus on a work of Tao Calligraphy art, tracing the characters with their fingers while simultaneously listening to or singing/chanting (silently or aloud) the Tao Music or Song, which enables them to achieve deep concentration and relaxation during wakefulness.

The Tao Song "Greatest Love" consists of short, inspiring verses that are repeated, and is a beautiful way to lift and inspire peoples' hearts and help them to experience peace and calm. The song was professionally recorded and is available for study participants as a free distribution.

The investigators have already discussed the value of Tao art mindfulness meditations for improving depression, anxiety, pain, and health, and how this appears to contribute to numerous beneficial outcomes related to well-being by the Short Form 36-item (SF-36) questionnaire to measure quality of life and by the European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC Quality of Life Questionnaire (QLQ) C-30).

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and over with a primary diagnosis as one Unipolar depression according to International Classification of Diseases (ICD)-10 criteria is present and diagnosed by a licensed physician.
* Willingness and ability to comply with data collection requirements
* Submission of required documentation before entering the study, including informed consent and consent to release of information
* Willingness to allow their data to be used for research purposes and published as deemed fit (while conforming to all applicable privacy laws) by Sha Research Foundation
* Willingness to practice the daily mindfulness practices for at least 30 minutes and follow the study protocol

Exclusion Criteria:

* Not meeting any of the inclusion criteria
* Bipolar disorders, schizophrenia (psychosis)
* Treatment with highly potent neuroleptics
* Unwillingness to participate in data gathering
* Unable to follow the practice regimen, including the daily individual mindfulness practices for at least 30 minutes
* Pregnant or nursing. Participants who become pregnant during the study will be required to end their participation.
* Serious mental disorders (e.g., schizophrenia)
* There is no exclusion criteria placed upon potential subjects related to national origin, culture, ethnicity, race, sex, physical disability, sexual orientation, religion, or spiritual practices.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Quality of Life Scores on 36-item short-form Quality of Life Questionnaire (SF-36) at 6 weeks | From start of Mindfulness practices with Tao Art (Calligraphy and Song Greatest Love) and drinking energized water to end of practices at 6 weeks.
  Description:
  A 36-item short-form Quality of Life Questionnaire (SF-36) was constructed to survey health status. The investigators chosen the longer 36-item version to assess the impact of the Tao art mindfulness practice and drinking energized water on Quality of Life of participants with unipolar depression.
  The SF-36 includes one multi-item scale for eight health concepts:
  1. limitations in physical activities;
  2. limitations in social activities;
  3. limitations in usual role activities;
  4. bodily pain;
  5. general mental health (psychological distress and well-being);
  6. limitations in usual role activities because of emotional problems;
  7. vitality (energy and fatigue);
  8. general health perceptions.
  Through a complex calculation, eight scores are derived from answers to 36 questions of SF-36. Finally, these eight scores are linearly transformed to a 0-to-100 scale, with 100 being the best possible outcome.
Mean Change from Baseline in Scores on PHQ-9 questionnaire at 6 weeks | From start of Mindfulness practices with Tao Art (Calligraphy and Song Greatest Love) and drinking energized water to end of practices at 6 weeks.
  The PHQ-9 questionnaire that measures criteria of Mental Disorders, will be used to assess the impact of the Tao art mindfulness practice and drinking energized water on unipolar depression.
  PHQ-9 has 9 scores, derived from answers to 9 questions of PHQ-9. These 9 scores have a 0-to-3 scale, with 3 being the worst possible outcome. Participants select the scale to each score depending on how frequently experience depressive symptoms during two weeks as: Not at all = 0; Several days = 1; More then half of the days = 2; Nearly every day = 3.
  Then, add up the scores for each item to get a total. Total scores on the PHQ-9 can range from 1 to 27, with higher scores indicating more severe Depression:
  * Scores ranging from 1-4 = minimal depression.
  * Scores ranging from 5-9 = mild depression.
  * Scores ranging from 10-14 = moderate depression.
  * Scores ranging from 15-19 = moderately severe depression.
  * Scores ranging from 20-27 = severe depression.
Mean Change from Baseline in Scores on BAI-21 (Beck Anxiety Inventory) Scale at 6 weeks | From start of Mindfulness practices with Tao Art (Calligraphy and Song Greatest Love) and drinking energized water to end of practices at 6 weeks.
  The BAI-21, Beck Anxiety Inventory Scale, will be used to assess the impact of the Tao art mindfulness practice and drinking energized water on unipolar depression.
  Each of the 21 items of BAI-21 is descriptive of subjective, somatic, or pain-related symptoms of anxiety. The participant rates how much he or she has been bothered by that symptom in the past week. Each question has the same set of four possible answer choices with a scale of 0-3, with 3 being the worst possible outcome.
  Then, add up the scores for each item to get a total. Total scores on the BAI-21 can range from 1 to 63, with higher scores indicating more severe Depression:
  * Scores ranging from 1-10 = normal ups and downs.
  * Scores ranging from 11-16 = mild mood disturbance.
  * Scores ranging from 17-20 = borderline depression.
  * Scores ranging from 21-30 = moderate depression.
  * Scores ranging from 31-40 = severe depression.
  * Scores ranging from 40-63 = extreme depression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hudoba De Badyn, MD, FRCS,, Principal Investigator — Sha Research Foundation; Laurie Omuro-Yamamoto, PhD, Principal Investigator — Satori Family Wellness Center
Locations (1):
- Satori Family Wellness Center, Kahului, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share the protocol with the statistical analysis plan of the study, the mean change from baseline in the SF-36 Quality of Life Scores, the PHQ-9 Patient Health Questionnaire Scores and the BAI-21 Beckman Anxiety Inventory Scores after six weeks of mindfulness practices with Tao Art and energized water.
Supporting Information: Study Protocol, SAP
Time Frame: The protocol with the statistical analysis plan of the study will be available from April 30, 2025 until the end of the study on January 10, 2027.
  The mean change from baseline in the SF-36 Quality of Life Scores, the PHQ-9 Scores and the BAI-21 Beckman Anxiety Inventory Scores after six weeks of mindfulness practices with Tao Art and energized water will be available from January 10, 2027 until December 31, 2027.
Access Criteria: Anyone with an active account at this platform.

REFERENCES:
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Kao HS, Lam SP, Kao TT. Chinese calligraphy handwriting (CCH): a case of rehabilitative awakening of a coma patient after stroke. Neuropsychiatr Dis Treat. 2018 Jan 31;14:407-417. doi: 10.2147/NDT.S147753. eCollection 2018. PMID 29440902
- [Result] Kobau R, Seligman ME, Peterson C, Diener E, Zack MM, Chapman D, Thompson W. Mental health promotion in public health: perspectives and strategies from positive psychology. Am J Public Health. 2011 Aug;101(8):e1-9. doi: 10.2105/AJPH.2010.300083. Epub 2011 Jun 16. PMID 21680918
- [Result] White JD. National Cancer Institute's support of research to further integrative oncology practice. J Natl Cancer Inst Monogr. 2014 Nov;2014(50):286-7. doi: 10.1093/jncimonographs/lgu036. No abstract available. PMID 25749590
- [Result] Marikar Bawa FL, Mercer SW, Sutton JW, Bond CM. Mindfulness for people with chronic pain: Factors affecting engagement and suggestions for programme optimisation. Health Expect. 2023 Jun;26(3):1287-1307. doi: 10.1111/hex.13745. Epub 2023 Mar 12. PMID 36908018
- [Result] Jamil A, Gutlapalli SD, Ali M, Oble MJP, Sonia SN, George S, Shahi SR, Ali Z, Abaza A, Mohammed L. Meditation and Its Mental and Physical Health Benefits in 2023. Cureus. 2023 Jun 19;15(6):e40650. doi: 10.7759/cureus.40650. eCollection 2023 Jun. PMID 37476142
- [Result] Pascoe MC, de Manincor M, Tseberja J, Hallgren M, Baldwin PA, Parker AG. Psychobiological mechanisms underlying the mood benefits of meditation: A narrative review. Compr Psychoneuroendocrinol. 2021 Mar 10;6:100037. doi: 10.1016/j.cpnec.2021.100037. eCollection 2021 May. PMID 35757358
- [Result] Poissant H, Mendrek A, Talbot N, Khoury B, Nolan J. Behavioral and Cognitive Impacts of Mindfulness-Based Interventions on Adults with Attention-Deficit Hyperactivity Disorder: A Systematic Review. Behav Neurol. 2019 Apr 4;2019:5682050. doi: 10.1155/2019/5682050. eCollection 2019. PMID 31093302
- [Result] de Witte M, Orkibi H, Zarate R, Karkou V, Sajnani N, Malhotra B, Ho RTH, Kaimal G, Baker FA, Koch SC. From Therapeutic Factors to Mechanisms of Change in the Creative Arts Therapies: A Scoping Review. Front Psychol. 2021 Jul 15;12:678397. doi: 10.3389/fpsyg.2021.678397. eCollection 2021. PMID 34366998
- [Result] de Witte M, Lindelauf E, Moonen X, Stams GJ, van Hooren S. Music Therapy Interventions for Stress Reduction in Adults With Mild Intellectual Disabilities: Perspectives From Clinical Practice. Front Psychol. 2020 Dec 10;11:572549. doi: 10.3389/fpsyg.2020.572549. eCollection 2020. PMID 33362637
- [Result] Kao H Sr, Zhu L, Chao AA, Chen HY, Liu IC, Zhang M. Calligraphy and meditation for stress reduction: an experimental comparison. Psychol Res Behav Manag. 2014 Feb 13;7:47-52. doi: 10.2147/PRBM.S55743. eCollection 2014. PMID 24611024
- [Result] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Result] Simpson FM, Perry G, Thompson WF. Assessing Vocal Chanting as an Online Psychosocial Intervention. Front Psychol. 2021 Jun 1;12:647632. doi: 10.3389/fpsyg.2021.647632. eCollection 2021. PMID 34140914
- [Result] Perry G, Polito V, Sankaran N, Thompson WF. How Chanting Relates to Cognitive Function, Altered States and Quality of Life. Brain Sci. 2022 Oct 27;12(11):1456. doi: 10.3390/brainsci12111456. PMID 36358382
- [Result] Spitzer RL, Williams JB, Kroenke K, Linzer M, deGruy FV 3rd, Hahn SR, Brody D, Johnson JG. Utility of a new procedure for diagnosing mental disorders in primary care. The PRIME-MD 1000 study. JAMA. 1994 Dec 14;272(22):1749-56. PMID 7966923
- [Result] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Result] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Result] Al Ozairi A, Alsaeed D, Al-Ozairi E, Irshad M, Crane RS, Almoula A. Effectiveness of virtual mindfulness-based interventions on perceived anxiety and depression of physicians during the COVID-19 pandemic: A pre-post experimental study. Front Psychiatry. 2023 Jan 9;13:1089147. doi: 10.3389/fpsyt.2022.1089147. eCollection 2022. PMID 36699484
- [Result] Trivedi MH. Major Depressive Disorder in Primary Care: Strategies for Identification. J Clin Psychiatry. 2020 Mar 17;81(2):UT17042BR1C. doi: 10.4088/JCP.UT17042BR1C. PMID 32220155
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Cassano P, Fava M. Depression and public health: an overview. J Psychosom Res. 2002 Oct;53(4):849-57. doi: 10.1016/s0022-3999(02)00304-5. PMID 12377293
- [Result] de Zwart PL, Jeronimus BF, de Jonge P. Empirical evidence for definitions of episode, remission, recovery, relapse and recurrence in depression: a systematic review. Epidemiol Psychiatr Sci. 2019 Oct;28(5):544-562. doi: 10.1017/S2045796018000227. Epub 2018 May 17. PMID 29769159
- [Result] Lee B, Wang Y, Carlson SA, Greenlund KJ, Lu H, Liu Y, Croft JB, Eke PI, Town M, Thomas CW. National, State-Level, and County-Level Prevalence Estimates of Adults Aged >/=18 Years Self-Reporting a Lifetime Diagnosis of Depression - United States, 2020. MMWR Morb Mortal Wkly Rep. 2023 Jun 16;72(24):644-650. doi: 10.15585/mmwr.mm7224a1. PMID 37318995

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT06934330/Prot_SAP_000.pdf